CLINICAL TRIAL: NCT03369301
Title: Effect of Subcutaneous Immunoglobulin (IgSC) Gammanorm® on the Distribution of IgG Subclasses and on the Humoral Immunity of Patients With Secondary Immunodeficiency.
Brief Title: The Effect of Subcutaneous Immunoglobulin Gammanorm on the Distribution of IgG Subclasses and on Immunity of Patients With Secondary Immunodeficiency
Status: Completed | Type: Observational
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Other Study IDs: Optinorm
Record Dates: First submitted 2017-11-30; First posted 2017-12-12 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Secondary Immune Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gammanorm: Patients on Gammanorm per standard of care
  Interventions: Drug: Gammanorm
- Other Subcutaneous Immunoglobulin: Patients on subcutaneous immunoglobulin treatments other than Gammanorm
  Interventions: Drug: Other Subcutaneous Immunoglobulins

INTERVENTIONS:
Drug: Gammanorm — Gammanorm given per standard of care
  Groups: Gammanorm
Drug: Other Subcutaneous Immunoglobulins — Other Subcutaneous Immunoglobulins given per standard of care
  Groups: Other Subcutaneous Immunoglobulin

SUMMARY:
Patients with Myeloma or CLL with severe secondary hypogammaglobinemia and recurrent infections will be included in this study; for whom an IgSC treatment was prescribed. The IgSC prescription will be the decision of the treating physician. Patient care and follow up will be performed according to the current clinical practice and the recommendations of HAS.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female (≥18 years old), Myeloma or Chronic Lymphocytic Leukemia patients with secondary hypogammaglobinemia and recurring infections.
2. Patients with indication for IgSC treatment but who have not started the treatment yet. Prior IgSC or IgIV treatment 6 months before inclusion is accepted (with a washout period of 6 months minimum).
3. Patient having received all the necessary information about the study and signed an informed consent document.

Exclusion Criteria:

1. Patient having initiated an IgSC treatment.
2. Patient having received IgSC or IgIV treatment within 6 months prior to inclusion.
3. Incapacity/Inability to attend the follow-up visits.
4. Patient refusing to participate in the study.
5. HIV positive patients.
6. Incapacity to understand the study objective and process, to agree or to give informed consent to participate in the study.
7. Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every eligible patient for the selection criteria will be consecutively included in the study to avoid any selection bias.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Distribution of difference subclasses of IgGs with respect to subcutaneous immunoglobulin treatment | 12 months
  Distribution of difference subclasses of IgGs with respect to subcutaneous immunoglobulin treatment collected as biological data including immunoglobulins (quantitative dosage and electrophoresis), lymphocytes, CD14 monocytes, polynuclear neutrophils, polynuclear basophils and dendritic cells

SECONDARY OUTCOMES:
Change in immune system | 12 months
  To analyze the change in the immune system (CD14 monocytes, polynuclear neutrophils, polynuclear basophils and dendritic cells)
IgG levels | 12 months
  To analyze the IgG levels with respect to the IgSC treatment
Lymphocytic Repertoire analyzing the evolution of the lymphocytic repertoire (CD3, CD4, CD8, CD19, CD56, and CD27). | 12 months
  To analyze the evolution of the lymphocytic repertoire (CD3, CD4, CD8, CD19, CD56, and CD27).
IgSC treatment | 12 months
  To characterize the IgSC treatment duration and the patient management (observance, duration and reason of termination)
Bacterial Infections | 12 months
  To evaluate the severe and non-severe bacterial infection rates
Antibiotic Consumption | 12 months
  To evaluate the antibiotics consumption during the study
Hospitalizations due to infections | 12 months
  Evaluate the hospitalization rates due to infections
Safety of IgSCs to characterize the IgSCs safety, including the adverse events that are not considered to be related to the study treatment | 12 months
  To characterize the IgSCs safety, including the adverse events that are not considered to be related to the study treatment
Predictive Factors of Recurrent Infections | 12 months
  To characterize potential predictive factors or markers of recurrent infections despite of the Ig treatment by collecting information about infections at follow up visits, especially bacterial infections and their respective antibiotherapy

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CH William Morey Chalon-sur-Saône, Chalon-sur-Saône
  - CHD Vendée, La Roche-sur-Yon
  - CH la Rochelle - Hôpital Saint Louis, La Rochelle
  - CH Orléans, Orléans
  - CHU Bordeaux Centre François Magendie Hopital Haut -Lévêque, Pessac
  - CH Saint Malo, St-Malo

IPD SHARING:
Plan to Share IPD: Undecided